CLINICAL TRIAL: NCT03178695
Title: Autologous Platelet-Rich Plasma (PRP) Infusions and Biomarkers of Ovarian Rejuvenation and Aging Mitigation
Brief Title: Inovium Ovarian Rejuvenation Trials
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascendance Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 882388
Record Dates: First submitted 2017-04-19; First posted 2017-06-07 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Perimenopausal Disorder; Menopause; Menopause, Premature; Menopause Related Conditions; Menopause Premature Symptomatic; Menopause Premature Asymptomatic; Premature Ovarian Failure; Premature Ovarian Failure, Familial; Premature Ovarian Failure 2A; Premature Ovarian Failure 3; Premature Ovarian Failure 4; Premature Ovarian Failure 1; Premature Ovarian Failure 5; Premature Ovarian Failure 6; Premature Ovarian Failure 7; Premature Ovarian Failure 9; Premature Ovarian Failure 8; Infertility; Infertility, Female; Infertility Unexplained
Keywords: Infertility; Pregnancy; Menopause; Perimenopause; Premature Ovarian Failure
MeSH Terms: conditions — Menopause, Premature; Primary Ovarian Insufficiency; Premature ovarian failure, familial; Premature Ovarian Failure 2a; Premature Ovarian Failure 3; Ovarian Dysgenesis 2; Premature Ovarian Failure 5; Premature Ovarian Failure 6; Premature Ovarian Failure 7; Infertility; Infertility, Female

STUDY DESIGN:
Intervention Model Description: A study group receives the intervention, which is compared in terms of efficacy against a matched group of control patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment Group (Experimental): PRP is freshly isolated from patients with diminished ovarian reserve as determined by at least one prior IVF cycle canceled for poor follicular recruitment response, or estimated by serum AMH and/or FSH, no menses for ≥1 year. Immediately following substrate isolation and activation with calcium gluconate, approximately 5 mL of autologous PRP is injected into each ovary under direct transvaginal sonogram guidance. AMH, FSH, and serum estradiol data will be recorded at 2wk intervals post-PRP and compared to baseline (pre-PRP) values.
  Interventions: Other: Autologous PRP injection into human ovarian tissue
- Comparison Group (No Intervention): Data collected from all patients in the Treatment Group will be compared to a dataset compiled from 25 - 50 women of similar age having received like treatment via IVF and gonadotropin stimulation for positive fertility outcomes in past clinical work at the Center for Advanced Genetics, as a comparison model and substitute control group. The purpose of this comparison will be to determine overall efficacy of the Inovium Ovarian Rejuvenation Treatment as separated from the standard efficacy rates of CAG-established IVF processes and gonadotropins used in the trial.

INTERVENTIONS:
Other: Autologous PRP injection into human ovarian tissue — Using FDA-approved equipment, blood plasma is received from participant, isolated/enriched into PRP, and infused into the ovaries under transvaginal ultrasound guidance.
  Arms: Treatment Group

SUMMARY:
The Inovium Ovarian Rejuvenation Treatment is a PRP-based autologous treatment used in combination with a stimulated IVF sequence and Pre-Implantation Genetic Screening to treat infertility in women experiencing menopause, perimenopause, and premature ovarian failure.

DETAILED DESCRIPTION:
This research extends earlier work conducted by Inovium associates in Athens, Greece who demonstrated efficacy of intraovarian injection of autologous PRP for resumption of menses, hormone stabilization, and conception after IVF in multiple women following PRP+natural cycle IVF (i.e., without gonadotropin stimulation). The use of stimulation (gonadotropins) and targeted pre- and posttreatment hormone monitoring during this clinical trial aims to characterize more fully the transition from PRP dosing, embryogenesis, IVF and conception.

The current study seeks to describe how PRP works to rejuvenate immune system and ovarian stem cells, restore menses, provide hormone stability, and generate successful IVF sequences and conceptions. The quality of all embryos generated will be studied via PGS, with the goal of generating euploid embryos. Hormone stability and biomarkers of aging will also be evaluated to understand the extent of any observed benefits, and to estimate how long such effects may be sustained with a single PRP treatment.

Autologous activated PRP used in this clinical study is isolated from patient derived (blood) samples collected on-site, using FDA-approved Regenlab [Lausanne, Switzerland] BCT-1 PRP Kit and RegenLab Drucker Centrifuge (FDA 510(k)-Approval #BK110061; ISO#13485).

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Women over the age of 35
* Primary or secondary amenorrhea at least for 3-6 months
* Presence of at least one ovary
* Agree to report any pregnancy to the research staff immediately.
* Willing and able to comply with study requirements.
* Willing to receive IVF to get pregnant as part of the experimental protocol.

Exclusion Criteria:

* Men will be excluded from the study.
* Current or previous IgA deficiency
* Current or previous premature ovarian failure due to a genetic origin, such as Turner's Syndrome or chromosomal abnormality
* Current or previous great injuries or adhesions to the pelvis or ovaries
* Current and ongoing pregnancy
* Current and ongoing anticoagulant use for which plasma infusion appears contraindicated
* Current and ongoing major Mental health disorder that precludes participation in the study
* Current and ongoing active substance abuse or dependence
* Current and ongoing gynecological or non-gynecological cancer
* Current and ongoing chronic pelvic pain

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Men are not eligible to participate in the trials.
Enrollment: 200 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Positive IVF | 12 months
  Following the initial Ovarian Rejuvenation Treatment, subjects will undergo IVF treatment to test the efficacy of the Protocol for fertility outcomes, as per trial protocols.
Positive Pregnancy and Conception | 12 months
  Following completion of trial protocols, patients will conduct ongoing post-treatment follow-up with trial staff for recording progress of all ongoing pregnancies and conceptions, via post-treatment correspondence.

SECONDARY OUTCOMES:
Resumption of Menses | 12 months
  With Premature Ovarian Failure and natural menopause the normal menstrual cycle is disrupted and normal menses does not occur. Patients will monitor for resumption of menses.
Changes in Hormone Levels | 12 months
  Changes in hormonal levels toward normal ranges. Hormones may include FSH/LH; Estradiol/ progesterone;Inhibin; Anti- Mullerian Hormone
Changes in Egg Quality | 12 months
  Using Pre-Implantation Genetic Screening, the trials will study the changes to egg quality of all eggs generated as a result of the treatment. A comparison group of patients who have received standard IVF treatment without the Inovium Ovarian Rejuvenation Treatment will be used to study this outcome.
Changes in Health Outcomes | 12 months
  Changes in overall health levels will be studied. A comparison group of patients who have received standard IVF treatment without the Inovium Ovarian Rejuvenation Treatment will be used to study this outcome. All patient data collected as described in the other outcomes will be used in this comparison.
Duration of Identified Benefits of Treatment | 12 months
  The duration of effects will be studied, in order to identify a frequency of treatment necessary to sustain positive health and fertility outcomes.
Changes in Menopausal Symptoms | 12 months
  A before-and-after questionnaire will be administered to collect patient personal experience data regarding changes in menopausal symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: E Scott Sills, MD PhD, Principal Investigator — Center for Advanced Genetics (CAG)
Locations (1):
- Center for Advanced Genetics, Carlsbad, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All requests and considerations for data sharing with individual and institutional researchers will be reviewed by the members of the Inovium Trials' Scientific Advisory Board and Primary Investigator.

REFERENCES:
- [Result] Sills ES, Rickers NS, Petersen JL, Li X, Wood SH. Regenerative effect of intraovarian injection of activated autologous platelet rich plasma: Serum anti-Mullerian hormone levels measured among poor-prognosis in vitro fertilization patients. International Journal of Regenerative Medicine 2020;3(1):1-5. https://www.sciencerepository.org/regenerative-effect-of-intraovarian-injection_RGM-2020-1-102
- [Result] Sills ES, Li X, Rickers NS, Wood SH, Palermo GD. Metabolic and neurobehavioral response following intraovarian administration of autologous activated platelet rich plasma: First qualitative data. Neuro Endocrinol Lett. 2019 Jan;39(6):427-433. PMID 30796792
- [Result] Sills ES, Rickers NS, Li X, Palermo GD. First data on in vitro fertilization and blastocyst formation after intraovarian injection of calcium gluconate-activated autologous platelet rich plasma. Gynecol Endocrinol. 2018 Sep;34(9):756-760. doi: 10.1080/09513590.2018.1445219. Epub 2018 Feb 28. PMID 29486615
- [Result] Sills ES, Rickers NS, Svid CS, Rickers JM, Wood SH. Normalized Ploidy Following 20 Consecutive Blastocysts with Chromosomal Error: Healthy 46, XY Pregnancy with IVF after Intraovarian Injection of Autologous Enriched Platelet-derived Growth Factors. Int J Mol Cell Med. 2019 Winter;8(1):84-90. doi: 10.22088/IJMCM.BUMS.8.1.84. Epub 2019 May 15. PMID 32195207
- See also: Clinical data (published) — https://www.sciencerepository.org/regenerative-effect-of-intraovarian-injection_RGM-2020-1-102